CLINICAL TRIAL: NCT01538082
Title: Role of Anxiety, Depression, Quality of Life and Stressful Vital Events in the Development of the Metabolic Syndrome. StreX Project.
Brief Title: Role of the Stress in the Development of the Metabolic Syndrome
Acronym: STREX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Societat Catalana de Medicina Familiar i Comunitària, Assoc. (CAMFiC) (Other); Spanish Society of Family and Community Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 7Z08/002
Record Dates: First submitted 2012-02-19; First posted 2012-02-23 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Anxiety Disorders; Depressive Disorders; Metabolic Syndrome; Stress Disorders
Keywords: Anxiety disorders; Depressive disorders; Metabolic syndrome; Stress disorders; Primary care
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder; Metabolic Syndrome; Stress Disorders, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients without stress: Patients without any of the next items: Zung's questionnaire score over 19 points; SF-12 questionnaire score over 5 points; Stressful vital events score over 150 points.
- Patients with stress: Patients with stress, including: Zung's questionnaire punctuation over 19 points; SF-12 questionnaire score over 5 points; stressful vital events score over 150 points. All combinations are considered positive in stress.

SUMMARY:
The purpose of this study is determine the incidence of metabolic syndrome (MetS) in people of high risk, of 40 or more years and attended in the Primary Care. Evaluating the association between anxiety, depression, quality of life and the vital stressful events, and the development of the metabolic syndrome in general population.

Our hypothesis is that population of the cohort with bigger degree of stress will develop earlier the metabolic syndrome.

If our hypothesis about the metabolic syndrome are demonstrated, it would allow establishing in a future interventions on these factors of risk to prevent or to decrease the incidence of this syndrome in the Primary Care.

ELIGIBILITY:
Inclusion Criteria:

* Both genders, elderly than 40 years
* Subjects with 1 or 2 criteria of NCEP-ATPIII set for Metabolic Syndrome

  * Abdominal waist > 102 cm ( men ) or >88 cm ( women )
  * Blood Pressure ( >130/85 mmHg ) ( or else pharmacologic treatment of hypertension )
  * Hypertriglyceridaemia ( >150 mg/dl ) ( or else pharmacologic treatment )
  * HDL-cholesterol <40 mg/dl ( men ) or <50 mg/dl ( women ) ( or else treatment )
  * Fasting glucose > 110 mg/dl.

Exclusion Criteria:

* Metabolic Syndrome (NCEP-ATPIII defined)(3 criteria of above mentioned)
* Severe or terminal disease
* Severe mental disease that difficulties the follow-up

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aleatory sample of subjects with high risk ( 1 or 2 criteria NCEP-ATPIII ) to develop Metabolic Syndrome, elderly than 40 years and attended in Primary Care in the last year. This sample will be provided by the Information's Technology in Primary Care Services.
Sampling Method: Probability Sample
Enrollment: 738 (Estimated)
Dates: Start 2008-12; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of metabolic syndrome | One year
  Determining the incidence of metabolic syndrome ( MetS ) in people of high risk, older than 40 years and attended in the Primary Care.

SECONDARY OUTCOMES:
Association between risk factors and metabolic syndrome | One year
  Association between anxiety, the depression, the quality of life and the vital stressful events and the metabolic syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Yolanda Ortega, MD, Principal Investigator — Catalan Institute of Health; Juan J Cabré, MD, PhD, Study Director — Catalan Institute of Health; Josep L Piñol, MD, PhD, Study Chair — Catalan Institute of Health
Locations (1):
- Catalan Health Institute. ABS Reus-4, Reus, Tarragona, Spain